CLINICAL TRIAL: NCT00772460
Title: Comparison of a New Patient Warming System Using Polymer Conductive Warming With Forced Air Warming During Surgery
Acronym: HDV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Dr. Oliver Kimberger, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HotDogVienna
Record Dates: First submitted 2008-10-14; First posted 2008-10-15 (Estimated); Last update posted 2009-09-21 (Estimated); Status verified 2009-09

CONDITIONS: Hypothermia
Keywords: patient warming; convective warming; conductive warming; intraoperative normothermia; accidental hypothermia; intraoperative hypothermia
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Forced Air (Active Comparator): Warming with forced air (BairHugger)
  Interventions: Device: Patient Warming with conductive / convective warming
- Conductive Warming (Experimental): Warming with the conductive device (HotDog)
  Interventions: Device: Patient Warming with conductive / convective warming

INTERVENTIONS:
Device: Patient Warming with conductive / convective warming — Warming device set to maximum (43 °C)

SUMMARY:
Two patient warming systems will be compared with 40 patients each in a convective warming group (BairHugger, Arizant) and in a conductive warming group (HotDog, Augustine Biomedical).

The patients will undergo small to medium trauma surgery and will be warmed with the randomized device - the hypothesis is, that the area under the standardized core temperature / time curve is significantly greater in the conductive warming group. Secondary outcome is the mean skin temperature / time area under the curve.

DETAILED DESCRIPTION:
General study design We will study 200 patients (18-90 years) undergoing elective orthopedic surgery at the trauma surgery unit. The patients must have normal weight (20-30 BMI), the duration of surgery should last between 3 - 4 hours. There will be no other exclusion criteria (except severe peripheral arterial disease in the warmed extremity), as forced air patient warming is routinely used for all patients during this procedure.

The patients will be randomly assigned via a computer generated randomization list to treatment with either polymer or forced air warming. Anaesthesia and fluid management will be administered as desired by the anaesthesiologist.

Before warming four skin temperature probes will be attached to the upper arm, chest, abdomen and back of the patients to calculate mean body temperature. A probe (Mallinckrodt Anesthesiology Products, Inc., St. Louis, MO) will be introduced in the ear to measure core temperature. Afterwards, treatment with BairHugger or HotDog will be started.

The measurements will be recorded every five minutes until the end of surgery when intraoperative warming is stopped.

Differences between core temperatures will be analyzed both by using the summary measure of AUC (area under the curve) and by comparing the core-temperature at the end of surgery in the polymer and the forced air group with two-tailed, unpaired t tests if normally distributed and with a Wilcoxon test, if not normally distributed (distribution tested by K-S-test).

Results are expressed as means ± standard deviations if normally distributed, as median (IQ-Range) when not normally distributed.

Differences will be considered statistically significant when P < 0.05. We consider a difference in core temperature at the end of surgery of 0.5°C as clinically important. Considering this difference as well as a known standard deviation of approximately 1.5°C we will have to study 40 patients in each arm of the study to achieve statistical significance using a power of 90% and a p-value of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* The patients must have normal weight (20-30 BMI), the duration of surgery should last between 3 - 4 hours.
* There will be no other exclusion criteria , as forced air patient warming is routinely used for all patients during this procedure.

Exclusion Criteria:

* Severe peripheral artery disease in the warmed extremity

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2008-10; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Area under the standardized "core temperature * time" curve | intraoperatively

SECONDARY OUTCOMES:
Area under "mean skin temperature * time" curve | intraoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Kimberger, M.D., Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Vienna, Austria

REFERENCES:
- [Derived] Brandt S, Oguz R, Huttner H, Waglechner G, Chiari A, Greif R, Kurz A, Kimberger O. Resistive-polymer versus forced-air warming: comparable efficacy in orthopedic patients. Anesth Analg. 2010 Mar 1;110(3):834-8. doi: 10.1213/ANE.0b013e3181cb3f5f. Epub 2009 Dec 30. PMID 20042442